CLINICAL TRIAL: NCT04896359
Title: Effect of High Doses of Vitamin C on the Tissular Reparation (Healing) in Patients Under Surgery in the "Hospital de Los Valles".
Brief Title: High Doses Vitamin C and Tissular Repair in Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Francisco de Quito (Other)
Collaborators: Biomolec Pharma (Unknown)
Responsible Party: Principal Investigator, Enrique Teran, Principal Investigator, Universidad San Francisco de Quito
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HUBI - 14539
Record Dates: First submitted 2021-05-11; First posted 2021-05-21 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Tissue Damage
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): i.v. infusion of 12.5 g vitamin C 48 h before surgery, immediately before surgery, and 48 h after surgery
  Interventions: Dietary Supplement: Vitamin C
- Control (Placebo Comparator): i.v. infusion of placebo 48 h before surgery, immediately before surgery, and 48 h after surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — 12.5 grams of ascorbic acid
  Arms: Vitamin C
Other: Placebo — vehicle
  Arms: Control

SUMMARY:
This is a prospective, randomize, double-blind, and placebo-controlled study to evaluate in patients with clinical criteria for any of the following open surgical procedure: (1) cesarean section; (2) aesthetic surgery like abdominoplasty; (3) orthopedic surgery; and (4) abdominal open surgery [excluding laparoscopic procedures] will be invited to receive either a high dose of vitamin C (12.5 g) three times (48 h pre-surgery, immediately before surgery and 48 h post-surgery) or its placebo, to evaluate the tissue repair process using an international validated instrument named Patient and Observer Scar Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Susceptible for any of the following surgical procedures: (1) cesarean section; (2) aesthetic abdominal plastic surgery; (3) orthopedic prosthetic replacement surgery
* Voluntary consent to participate

Exclusion Criteria:

* Known allergy to the vitamin C
* Known problems with wounds healing
* Kidney disease (including lithiasis) or gout

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of linear scars | initial assessment, two weeks after surgery
  Patient and Observer Scar Assessment Scale (it evaluates in a 0 to 10 scale: vascularity, pigmentation, thickness, relief, pliability and surface area)
Evaluation of linear scars | second assessment, one month after surgery
  Patient and Observer Scar Assessment Scale (it evaluates in a 0 to 10 scale: vascularity, pigmentation, thickness, relief, pliability and surface area)
Evaluation of linear scars | third assessment, three months after surgery
  Patient and Observer Scar Assessment Scale (it evaluates in a 0 to 10 scale: vascularity, pigmentation, thickness, relief, pliability and surface area)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Teran, Principal Investigator — Universidad San Francisco de Quito
Locations (1):
- Hospital de los Valles, Quito, Pichincha, Ecuador